CLINICAL TRIAL: NCT05536063
Title: Effect of Dexamethasone as an Adjuvant to Bupivacaine in Bilateral Erector Spinae Block on Postoperative Pain and Diaphragmatic Function After Pediatric Cardiac Surgeries : A Randomized Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amonios khalil, assistant lecturer at anaesthesia and ICU department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESPB in ped. cardiac surgeries
Record Dates: First submitted 2022-08-23; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Pediatric Cardiac Surgery

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Experimental): bilateral ESPB with 0.5 ml/kg of 0.25% bupivacaine (limited to a maximum dose of 20 ml) for each side
  Interventions: Procedure: bilateral erector spinae plane block in pediatric cardiac surgeries
- Group B (Experimental): bilateral ESPB with 0.5 ml/kg of 0.25% bupivacaine (limited to a maximum dose of 20 ml) + dexamethasone 0.1 mg/kg for each side
  Interventions: Procedure: bilateral erector spinae plane block in pediatric cardiac surgeries
- Group C (No Intervention): control group will receive the standard analgesic regimen only

INTERVENTIONS:
Procedure: bilateral erector spinae plane block in pediatric cardiac surgeries — The ESPB will be performed after induction of anesthesia, endotracheal tube insertion and before the start of operation, with the child in a right lateral decubitus position under aseptic precautions. A high frequency linear ultrasound transducer will be placed over the T4 transverse process lateral to the spinous process. After identifying the muscles above the hyperechoic transverse process image, a 5-cm 22 gauge needle will be inserted in-plane in a cephalo-caudad direction. The endpoint is defined as the needle pointing to the tip of transverse process piercing the erector spinae muscle. The local anesthetic will be deposited at this position, After careful negative aspiration, local anesthetic, according to study groups , The process will be repeated on thecontralateral side
  Arms: Group B; group A

SUMMARY:
The aim of this study is to figure out the efficacy of dexamethasone addition to bupivacaine versus bupivacaine alone in bilateral erector spinae plane block on postoperative analgesia after pediatric cardiac surgeries

DETAILED DESCRIPTION:
The recently introduced ultrasound-guided interfascial plane block, bilateral erector spinae plane block (ESPB) is a viable option for management of postoperative pain after midline sternotomy. It is expected to provide an analgesic cover spanning the entire thorax at the desired dermatomes including the midline, which could prove beneficial for cardiac surgery through midline sternotomy.

Indications for ESPB for postoperative analgesia in pediatric surgeries to date include thoracotomy, video-assisted thoracoscopic surgery, vascular ring repair and sternotomy.

Dexamethasone is a synthetic glucocorticoid acting as an anti- inflammatory. It inhibits the release of inflammatory mediators such as interleukins and cytokines. Several studies have shown that a preoperative dose of dexamethasone added to local anesthetic agents has promising results in reducing postoperative pain and improving the quality of analgesia

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I and II
* Undergoing cardiac surgical procedures through a midline sternotomyPreoperative ejection fraction <35%

Exclusion Criteria:

* Low-cardiac-output syndrome
* Ventricular arrhythmia
* Preoperative inotropic support
* Known allergies to any of the study drugs
* Intubation for more than 3 hours or re-exploration
* A redo or emergency surgery
* Contraindications to regional anesthesia as coagulopathy and infection in site of block.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
postoperative pain, Face, Legs, Activity, Cry and Consolability (FLACC) pain scale | Postoperative pain assessment is performed using FLACC pain scale at fixed time intervasl for 48 hours post extubation,
  The primary outcome of this study is the intensity of postoperative pain that will be assessed using Face, Legs, Activity, Cry and Consolability, minimum value 0 and maximum value 10, high scores means worse outcome (FLACC) pain scale

SECONDARY OUTCOMES:
total analgesic consumption postoperative | for 48 hours postextubation
  total amount of postoperative analgesic consumption

OTHER OUTCOMES:
Beta endorphins levels | Blood samples for postoperative beta-endorphins at 2, 24, and 48 hours post-extubation
  comparison between preoperative and postoperative levels of B-endorphins

REFERENCES:
- [Background] Karacaer F, Biricik E, Ilginel M, Tunay D, Topcuoglu S, Unlugenc H. Bilateral erector spinae plane blocks in children undergoing cardiac surgery: A randomized, controlled study. J Clin Anesth. 2022 Sep;80:110797. doi: 10.1016/j.jclinane.2022.110797. Epub 2022 Apr 28. PMID 35489304
- [Background] Ferrari G, De Filippi G, Elia F, Panero F, Volpicelli G, Apra F. Diaphragm ultrasound as a new index of discontinuation from mechanical ventilation. Crit Ultrasound J. 2014 Jun 7;6(1):8. doi: 10.1186/2036-7902-6-8. eCollection 2014. PMID 24949192